CLINICAL TRIAL: NCT05792917
Title: Bioequivalence Study of Tafolecimab Injections Manufactured by Two Different Processes in Chinese Healthy Male Volunteers
Brief Title: Bioequivalence Study of Tafolecimab Injections in Chinese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CIBI306K101
Record Dates: First submitted 2023-03-06; First posted 2023-03-31 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tafolecimab (a modified manufacturing process) (Experimental): 450mg，SC，single dose
  Interventions: Drug: tafolecimab (a modified manufacturing process)
- tafolecimab (a original manufacturing process) (Active Comparator): 450mg，SC，single dose
  Interventions: Drug: tafolecimab (a original manufacturing process)

INTERVENTIONS:
Drug: tafolecimab (a modified manufacturing process) — 450mg，SC，single dose
  Other Names: IBI306 (a modified manufacturing process)
  Arms: tafolecimab (a modified manufacturing process)
Drug: tafolecimab (a original manufacturing process) — 450mg，SC，single dose
  Other Names: IBI306 (a original manufacturing process)
  Arms: tafolecimab (a original manufacturing process)

SUMMARY:
This trial is conducted in China. The purpose of this study is to evaluate the pharmacokinetic similarity of Tafolecimab with different manufacturing process in healthy male subjects. Another purpose is to determine safety, and immunogenicity of sintilimab with different manufacturing process,also to determine Pharmacodynamics of Tafolecimab with different manufacturing process

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between 18 and 65 years of age, inclusive.
2. Low-density lipoprotein cholesterol (LDL-C) within the range of 1.8 mmol/L to 4.9 mmol/L, inclusive, at screening.
3. Body weight within the range of 63.0 kilograms (kg) to 75.0 kg, inclusive.
4. Subjects who are willing maintain current normal diet and physical activity.
5. Subjects agree to use reliable contraceptive measures (such as abstinence, sterilization, contraceptives, injectable contraceptive medroxyprogesterone or subcutaneous implant contraception, etc.) during the study period and within 6 months after the study drug infusion.
6. No history of serious diseases, including (but not limited to) cardiovascular, hepatic, renal, gastrointestinal, psychiatric, neurologic, endocrine, pulmonary, hematological, immune disease.
7. Subjects voluntarily signed the informed consent form and agreed to strictly follow the requirements of this protocol.

Exclusion Criteria:

1. Subjects who have a history of allergy, or may be allergic to the investigational drug and the related compounds.
2. Have used the inhibitors of proprotein convertase subtilisin type 9 (PCSK-9).
3. Have clinically relevant abnormalities identified by Vital signs, physical examination, clinical laboratory tests, 12-lead ECG, or chest X-ray, at screening.
4. Unwilling to stop any strenuous physical activity (such as weightlifting or long-distance running) within 72 hours before the planned follow-up visit.
5. History of hospitalization within 1 month before screening, major surgery within 6 months before screening, or other unstable conditions judged by the investigator.
6. The last dose of the previous investigational product which is chemical drug has been given in less than 1 month before administration.
7. The last dose of the previous investigational product which is biological drug has been given in less than 3 months before administration.
8. Have used any drugs (including over-the-counter drugs or prescription drugs), the last medication is less than 14 days or the last medication is less than 5 half-lives of the drug from the administration day (whichever is longer), or are using any drugs.
9. Have used any traditional Chinese medicines, vitamins or drugs or supplements known to affect lipid metabolism within 30 days before administration.
10. Have a positive test result of human immunodeficiency virus (Human Immunodeficiency Virus, HIV) antibody, hepatitis B virus surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or syphilis test at screening.
11. History of alcohol or drug abuse results within 12 months before screening. Average daily alcohol intake is more than 3 units of alcohol (male) (1 unit≈360mL beer, or 45mL spirits with 40% alcohol content, or 150mL wine), or unwilling to stop drinking 72 hours before administration and throughout the study period, or a positive ethanol breath test at screening, or positive drug screening results by urine at screening.
12. unable to abstain from smoking, alcohol and caffeinated beverages within 72 hours before administration and throughout the study period.
13. lost blood, donated blood ≥200 ml within 2 months before screening.
14. History of organ transplantation or malignant tumor.
15. Not suitable for this study in the investigator's opinion.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence results using the peak serum drug concentration (Cmax) as the judging indicators | up to Day 57
Bioequivalence results using the area under the serum concentration-time curve (AUC0-inf) as the judging indicators | up to Day 57

SECONDARY OUTCOMES:
Other PK parameters: Area under the plasma concentration-time curve (AUClast) | up to Day 57
Other PK parameters: Volume of distribution (V) | up to Day 57
Other PK parameters: elimination half-life (t1/2) | up to Day 57
Number of participants with adverse events, with abnormal vital signs, abnormal physical examination, abnormal laboratory test results and abnormal ECG readings | up to Day 57
The occurrence of Anti-drug Antibody(ADA) | up to Day 57
The occurrence of Neutralizing antibodies Antibody(NAb) | up to Day 57
Percentage Change from baseline in Low Density Lipoprotein choleterol (LDL-C) | up to Day 57
Percentage Change from baseline in Proprotein convertase subtilisin/kexin type 9(PCSK-9) | up to Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No